CLINICAL TRIAL: NCT00806104
Title: Effect of Dietary Supplementation With Fructo-oligosaccharides on Visceral Sensitivity and on Taxonomic and Functional Composition of Intestinal Microbiota of IBS Patients
Brief Title: Fructo-oligosaccharides and Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beghin-Meiji (Industry)
Responsible Party: Frederique Respondek / Scientific Affairs Manager, Beghin Meiji
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: FOS_QLV2
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — fructooligosaccharide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Fructo-oligosaccharides
  Interventions: Dietary Supplement: Fructo-oligosaccharides
- 2 (Placebo Comparator): Maltodextrins
  Interventions: Dietary Supplement: Maltodextrins

INTERVENTIONS:
Dietary Supplement: Fructo-oligosaccharides — Dietary supplementation for 4 weeks
  Arms: 1
Dietary Supplement: Maltodextrins — Dietary supplementation for 4 weeks
  Arms: 2

SUMMARY:
Fructo-oligosaccharides are known as prebiotic ingredients to modulate the composition of the intestinal microbiota and particularly to stimulate the growth of Bifidobacteria. Imbalance of the intestinal microbiota such as reduction of Bifidobacteria is implicated in Irritable Bowel Syndrome (IBS). Thus the objective of the study is to evaluate the effect of fructo-oligosaccharides to improve IBS score and to explore which modifications of the microbiota are responsible of this improvement.

ELIGIBILITY:
Inclusion Criteria:

* IBS subjects according to Rome III criteria
* Incomfort below or equivalent to 30mmHg during Tensostat test
* between 18 and 60 years
* no antibiotic treatment for the last 2 months
* less than 20g of dietary fibres consummed per day
* no analgesic treatment
* no treatment for intestinal transit

Exclusion Criteria:

* subjects suffering from diabetes, colic cancer, inflammatory bowel disease, dysthyroidy, Hirschprung disease, anorexia
* excessive consumption of alcohol or tobacco
* participating to another clinical study
* pregnant women
* antidepressor or anxiolytic treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
rectal sensitivity | 4 weeks

SECONDARY OUTCOMES:
taxonomic composition of intestinal microbiota | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michel Dapoigny, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- CHU Clermont Ferrand, Clermont-Ferrand, France
- Vall Hebron Hospital, Barcelona, Spain